CLINICAL TRIAL: NCT00709540
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacodynamics of ACE-011 (ActRIIA-IgG1) in Healthy Postmenopausal Women
Brief Title: A Safety, Tolerability and Pharmacodynamics Study of ACE-011 (ActRIIA-IgG1) in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A011-02
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single (Experimental): 10 subjects (8 active and 2 placebo)
  Interventions: Biological: ACE-011 or placebo

INTERVENTIONS:
Biological: ACE-011 or placebo — multiple administrations of ACE-011 given subcutaneously once per month for 3 months (4 administrations total)

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-dose, dose-escalating study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ACE-011 in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a postmenopausal woman, 45-85 years old (inclusive).
2. Subject has had 12 months of spontaneous amenorrhea, OR 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels >40 IU/L OR is 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
3. Subject is taking at least 500 mg of calcium supplement and 400 IU of vitamin D daily and has been following this regimen for at least 4 weeks prior to the first dose of study drug administration.
4. Subject has a body mass index (BMI) of ≥ 18.5 to < 30.
5. Subject must give written informed consent. If required by local law, candidates must also authorize the release and use of protected health information (PHI).

Exclusion Criteria:

1. Subject has a history of clinically significant major disease (as determined by the Investigator).
2. Subject has a history of hyperparathyroidism, hypoparathyroidism, hypocalcemia, rheumatoid arthritis, myeloproliferative disorder, gout, Paget's disease of the bone, or osteomalacia.
3. Subject has had a long bone fracture within the past 6 months prior to enrollment, or an osteoporosis-related fracture within the previous 2 years.
4. Subject has a history of opportunistic infection, or has had a serious local or systemic infection within 3 months prior to screening.
5. Subject has a history of severe allergic or anaphylactic reactions.
6. Subject had major surgery within the previous 3 months.
7. Subject has a history of drug or alcohol abuse, or tests positive in a drug and alcohol screen at screening or on Day 1 prior to dosing.
8. Subject consumed any alcohol within 72 hours prior to dosing.
9. Subject gave a blood donation (one unit or more) within 1 month prior to dosing, or plans to give a blood donation during the course of the study.
10. Subject has taken any of the following bone active medications:

    * Teriparatide at any time in their lifetime.
    * Fluoride therapy for more than 3 months during the previous 2 years.
    * Estrogen, androgen, anabolic steroids, corticosteroids (excluding inhaled, topical or local injections for joint pain), calcitonin, or other bone active drugs (e.g. selective estrogen receptor modulators) within the 4 months prior to screening.

    Bisphosphonates:
    * If treated for more than 6 months at any time in their lifetime.
    * If treated for 3 to 6 months within 2 years of screening.
    * If treated for less than 3 months within 6 months of screening.
11. Subjects with chronic stable diseases including migraines, hypertension, hyperthyroid disorder, hypothyroid disorder, gastroesophageal reflux disease, or mild depression/anxiety will be excluded unless the investigator does not have safety or compliance concerns at study entry.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple, escalating doses of ACE-011 in healthy postmenopausal women. | specified timepoints in the protocol

SECONDARY OUTCOMES:
To estimate the pharmacokinetic (PK) parameters of multiple, escalating doses of ACE-011 administered subcutaneously and to determine the effect of ACE-011 on bone mineral density (BMD) and biochemical markers of bone formation and resorption. | at specified timepoints in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ababa, MD, Principal Investigator — West Coast Clinical Trials
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States